CLINICAL TRIAL: NCT00721149
Title: NAVISTAR® THERMOCOOL® Catheter for the Radiofrequency Ablation of Symptomatic Paroxysmal Atrial Fibrillation- Treatment Use Study
Acronym: AFTX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment stopped after CDRH Advisory Panel (Nov 20, 2008) recommended NAVISTAR® THERMOCOOL® catheter approval.
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BWI03130TXA
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Diseases; Arrhythmia; Atrial Fibrillation
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Ablation; Non-randomized
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NaviStar ThermoCool (Experimental)
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — The Biosense Webster® NAVISTAR THERMOCOOL Diagnostic/Ablation Deflectable Tip Catheter is a luminal catheter with a deflectable tip designed to facilitate electrophysiological mapping of the heart and to transmit radiofrequency current to the catheter tip electrode for ablation purposes.

SUMMARY:
This trial evaluates the safety and effectiveness of catheter ablation for PAF. The investigational catheter being studied is the NAVISTAR® THERMOCOOL® irrigated-tip catheter. At the time of this study, the NAVISTAR® THERMOCOOL® Catheter was FDA-approved for commercial distribution in the U.S. for treating patients with Type I atrial flutter and drug refractory monomorphic sustained ventricular tachycardia post myocardial infarction. The catheter was approved for use in Europe for endocardial ablation for treating cardiac arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic PAF who have had three (3) AF episodes in the six (6) months prior to enrollment, one of which must be documented. Documentation may include electrocardiogram (ECG), transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip.
* Failure of at least one AAD for PAF [class I or III or AV nodal blocking agents such as beta blockers (BB) and calcium channel blockers (CCB)] as evidenced by recurrent symptomatic PAF, or intolerable side effects due to AAD.
* Signed Patient Informed Consent Form.
* Age 18 years or older.
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non- cardiac cause.
* Previous ablation for atrial fibrillation.
* Patients on amiodarone therapy at any time during the previous six (6) months.
* AF episodes that last longer than 30 days and are terminated via cardioversion.
* Any valvular cardiac surgical procedure.
* CABG procedure within the last 180 days (six months).
* Awaiting cardiac transplantation or other cardiac surgery within the next 360 days (12 months).
* Documented left atrial thrombus on imaging (e.g. TEE).
* History of a documented thromboembolic event within the past one (1) year.
* Diagnosed atrial myxoma.
* Presence of implanted ICD.
* Significant pulmonary disease, (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
* Women who are pregnant (by history of menstrual period or pregnancy test if the history is considered unreliable).
* Acute illness or active systemic infection or sepsis.
* Unstable angina.
* Myocardial infarction within the previous 60 days (two months).
* LVEF < 40%.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation (i.e. heparin or warfarin).
* Contraindication to CT/MRA procedure.
* Life expectancy less than 360 days (12 months).
* Enrollment in an investigational study evaluating another device or drug.
* Uncontrolled heart failure or NYHA class III or IV heart failure.
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
* Presence of a condition that precludes vascular access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilber, MD, Principal Investigator — Loyola University Medical Center Chicago

RESULTS

PARTICIPANT FLOW:
Groups:
- NAVISTAR® THERMOCOOL® Catheter: The Biosense Webster NAVISTAR® THERMOCOOL® Diagnostic/Ablation Deflectable Tip Catheter is a luminal catheter with a deflectable tip designed to facilitate electrophysiological mapping of the heart and to transmit radiofrequency current to the catheter tip electrode for ablation purposes.
Period: Overall Study
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Started | 10 (Enrollment was stopped after 10 subjects entered the trial.)
Completed | 9
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Hypertension Condition [Number; unit: Participants]
  With Hypertension | 3
  Without Hypertension | 7
Atrial Flutter Condition [Number; unit: Participants]
  With Atrial Flutter | 2
  Without Atrial Flutter | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Exhibited no Documented Symptomatic Paroxysmal Atrial Fibrillation (PAF) Episodes From Study Day 91 Through Day 361.
Description: A subject who exhibited no documented symptomatic PAF episodes was one who 1) had 2 or fewer repeat ablations within 90 days of the initial ablation with investigational catheter; 2) had an addition of antiarrhythmic medication which was previously ineffective for atrial fibrillation and did not exceed the previous historical maximum dosage (24 hour total dose); 3) was on atrioventricular nodal blocking agents such as beta blockers and/or calcium channel blockers and might be maintained at the current dose (ie, did not exceed previous historical maximum dosage (24 hour total dose).
Time Frame: From study day 91 through day 361
Population: The subjects who had a study ablation procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 9
Percentage of participants | 66.7

2. Primary Outcome: The Percentage of Subjects Who Experienced Incidences of Early Onset (Within 7 Days of Ablation Procedure) Catheter-related Adverse Events.
Description: Catheter-related adverse events include death, myocardial infarction, pulmonary vein stenosis, diaphragmatic paralysis, atrio-esophageal fistula, transient ischemic attack, stroke, cerebrovascular accident, thromboembolism, pericarditis, cardiac tamponade, pericardial effusion, pneumothorax, atrial perforation, vascular access complications, pulmonary edema, hospitalization (initial and prolonged), and heart block.
Time Frame: within 7 days of ablation procedure
Population: The subjects who had a study ablation procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 9
Percentage of participants | 0.0

3. Secondary Outcome: Percentage of Subjects Who Achieved Acute Success
Description: Acute success is defined as the confirmation of entrance block in all targeted pulmonary veins. Acute failure is defined as subjects who have a non-investigational catheter used for ablation of any atrial fibrillation targets or subjects who undergo more than 2 repeat ablation procedures or an ablation procedure beyond day 90.
Time Frame: Day 91 - 361
Population: The subjects who had a study ablation procedure.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 9
Percentage of participants | 100

4. Secondary Outcome: 24-hour Holter Data
Time Frame: 1 year
Population: Data not analyzed due to study termination - insufficient data to identify meaningful differences and draw significant conclusions.
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 0

5. Secondary Outcome: TTM Data
Time Frame: 1 year
Population: as for outcome 4
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Subjects Who Responded to Quality of Life Assessment
Description: SF 36 Symptom Frequency and Severity Checklist
Time Frame: 1 year
Population: as for outcome 4
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | NAVISTAR® THERMOCOOL® Catheter
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVISTAR® THERMOCOOL® Catheter (N=9)
Small hematoma - left groin (Blood and lymphatic system disorders) | 1 (1)
Gallstone, pancreatitis, cholelithiasis (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Because of early study termination, the study did not reach its targeted enrollment and study data analysis was not fully conducted, thus study results may not be interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is allowed to publish but must submit draft publication(s) to Biosense Webster, Inc. at least 30 days prior to submission for publication or presentation.